CLINICAL TRIAL: NCT00920673
Title: Age Influence on the Modifications of the Oral, Pharyngeal and Laryngeal Axis Alignment in Children Induced by Head Extension: an MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/06; 2009-A00163-54
Record Dates: First submitted 2009-06-09; First posted 2009-06-15 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Head Extension on the Anatomic Axes of the Superior Airway
Keywords: child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MRI — MRI during 35 to 65 minutes

SUMMARY:
In pediatric anesthesia and in pediatric intensive care, tracheal intubation is one of the most important procedure. To achieve this procedure as fast as possible and in is best conditions, the physician should choose the head posture which a priori will enable at first the best glottic visualisation during laryngoscopy, and at second will facilitate the route of the tube from the larynx to the trachea.

Tracheal intubation is a procedure used for years, and many textbooks recommendations on the best head posture for tracheal intubation in paediatrics have been made. Briefly summarized, depending on the age of the child, the head should (or not) be slightly extended, and a pillow should (or not) be positioned under the occiput. These recommendations are questionable for three majors reasons:

* despite an apparent consensus, some recommendations are quite different.
* none are based on anatomical nor clinical studies
* if for all of them, the age of the child is considered as critical point, but children are only grossly categorized in three categories (newborn, infants and old children). And the clinician has no way, facing a child, to make his choice between dichotomic attitudes.

Actually, the responses to these questions should need rigourous clinical studies on laryngoscopy, hard to design and very difficult to make. P.Adnet et coll. (Anesthesiology 2001) showed that an anatomical study with resonance magnetic imaging (MRI) can bring indirect but strong evidence and can be a first step leading to clinical studies. Many children need MRI study for different reasons, and it is fast and easy to get during their examination additional images of the superior airway.

In their unit, the investigators are experienced in this kind of study, as they recently published (Pediatric Anesthesia 2008) an MRI study demonstrating that in children, head extension improves the alignment of the visualisation axis on the laryngeal axis, but worsens the alignment of the pharyngeal axis on the laryngeal axis. However, patients included in their study were in major part infants, so the influence of the age could not be properly analyzed. Morevover, this study suffered of two main limitations, the lack of standardisation of head postures, and that a laryngeal mask the children, who were on general anesthesia (required for the MRI examination) were made using a laryngeal mask (as it was at this time the standard in their institution).

The investigators propose an MRI study of the influence of age on the consequences of head extension on the anatomic axes of the superior airway in children, with a prospective stratified on age study. Several modifications and improvement in the design of this study would diminished the limitations of the first study.

ELIGIBILITY:
Inclusion Criteria:

* No obesity
* No macro- or micro-cephaly
* No facial dysmorphism
* No tumor near to the superior airway

Exclusion Criteria:

* Premature child
* MRI in emergency
* Discovery of a tumor near to the superior airway during the MRI

Ages: 42 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To study the influence of age on the consequences of head extension on the anatomic axes of the superior airway in children | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Vialet, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (2):
- France (2):
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - Assistance Publique-Hopitaux de Marseille, Marseille